CLINICAL TRIAL: NCT03473327
Title: Immunological and Oxidative Stress Response in Relation to Abdominal Cancer Surgery
Acronym: IMOX
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Sara Kehlet Watt, MD, Zealand University Hospital
Other Study IDs: IMOX
Record Dates: First submitted 2016-02-29; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal neoplasms; Immunologic Factors; Postoperative Period
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for Whole Blood genomic profiling
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to characterize the systemic stress response (SSR) induced in patients undergoing colorectal cancer (CRC) surgery. The project is a clinical prospective study. Blood samples will be collected from 30 patients on the day before CRC-surgery, and 1, 2, 3 and 10 days after surgery. A specimen from the resected tumor tissue will also be collected and sent for immunohistochemical analysis. Whole blood gene expression profiling will be performed to gain knowledge of the genetic changes in immunological, inflammatory and oxidative stress-related factors initiated by surgery. Peripheral immunological cells, proteins and cytokines will be analysed by FLOW and ELISA methods, and the functional capacity of NK-cells will also be defined for each time point. Furthermore, tumor tissue will be analyzed for invasion of immunological cells. At each time point, the patients will be asked to fill out a validated patient reported outcome measure with questions concerning clinical outcome parameters related to recovery after CRC-surgery

DETAILED DESCRIPTION:
Background

The perioperative period is relatively short, but highly critical for cancer related survival. The surgical procedure results in release of tumor cells locally and in the blood, and induction of a surgical stress response (SSR). This leads to paralysis of the immune system, reduced clearance of cancer cells and optimal conditions for cancer cells to grow and metastasize(1).

Colorectal cancer (CRC) is the third most common cause of cancer in Denmark. In 2013, 4196 Danish patients were diagnosed with CRC(2) and current standard of care includes a tumour resection. However, even after an expected curative surgical tumour resection, 25-30% will have a relapse within 5 years after the primary procedure.

To improve the outcome after surgery for cancer, it is crucial to understand, in details, how SSR affects the immune response and how SSR affects the ability of cancer cells to grow and metastasize. By performing expression profiling of over 40.000 genes in whole blood before and after surgery, we will obtain a genetic signature of genes from circulating immune cells, including granulocytes, monocytes, B and T cells, dendritic cells, and platelets, which will enable us to see the exact impact surgery has on gene transcription of these immunological factors. By using this information, perioperative interventions can be performed to optimize the immunological response in the perioperative period, leading to reduced risk of cancer recurrence and consequently improved survival (3).

Surgical stress response (SSR) It is well known that a surgical procedure induces a disturbance of the immunological and inflammatory balance, causing a systemic inflammatory response (4), immune suppression (4,5) and excess reactive oxygen species (ROS) (6,7). Systemic inflammation promotes tumor growth (8), and in patients who have undergone potentially curative resection for colorectal cancer, the presence of a systemic inflammatory response predicts a poor outcome (3). The paralysis of the immune system includes reduced activity of NK cells and macrophages, both of which under normal circumstances protects against metastasis by eliminating disseminating tumor cells. Excessive ROS causes DNA damage, break down of extracellular matrix and elimination of cell-cell adhesions (5,6,7). In this way, surgery promotes optimal conditions for cancer cells to grow and metastasize in the post-operative phase. Recent research shows that immune cells and their invasion of the primary tumor correlates to the patient's prognosis, again suggesting that the immune response is important for inhibition of cancer growth(9,10). Detailed information of genetic changes in different factors of the immune response due to surgery remains unclear.

Study design The project consist of a clinical prospective explorative study including 30 patients undergoing elective hemi-colectomy due to colon cancer UICC stadium II-III. Blood samples will be collected on the day prior to surgery, and on post-operative day 1, 2, 3 and 10. Samples will be prepared for Flow cytometric analysis, bio banking, cryopreservation and whole blood genomic profiling.

Whole blood gene expression profiling will be performed and analyzed to determine possible transcriptional changes in genes encoding for immunological, inflammatory and oxidative stress-related factors caused by surgery. It is possible to make both a quantitative as well as qualitative measurement of these genetic changes (11).The probe sets that are found to be the most significantly differentially expressed before and after surgery will be chosen for further analysis. Genes that are significantly deregulated and have been described in previous studies, within the field of inflammation, immunological and oxidative stress, will be chosen for further analysis. Examples of exact genes within immunology and inflammation will be genes encoding for TNFα, IL-1b, IL-2, IL-6, IL-10, VEGF, TGFβ and HLA-G. Within oxidative and antioxidative genes, special emphasis will be taken in FoxO3, TP53 and ATM as inactivation of these are associated with increased levels of ROS. Upregulation of ATOX1, DEFB122 and GBX8 is associated with increased levels of ROS, and will also be chosen for further analysis (19-21).

Alterations in specific inflammatory and immune modulating proteins (TNFα, IL-1b, IL-2, IL-6, IL-10, VEGF, TGFβ and HLA-G), the functional activity of natural killer (NK) cells, and the fractions and absolute numbers of specific sub-populations of immune cells (CD3+CD4+, CD3+CD8+, FoxP3+ / CD4+CD25+CD127 /dim regulatory T cells, CD4+HLA-G+ regulatory T cells, myeloid-derived suppressor cells and NK subsets) will be identified. Results from genetic transcription analysis and analysis of alterations in inflammatory and immune modulating proteins, will be compared in order to give a full overview of the SSR, and the effect of surgery on immunological, oxidative and inflammatory factors, in order to evaluate the potential carcinogenic effect of surgery, and times and methods of optimal intervention in this damaging process.

Tumor samples from the 30 enrolled patients will be analyzed for the level of invasion of immunological cells. The results will be correlated to the results from gene expression profiling and analysis of inflammatory and immune modulating proteins determined in whole blood samples prior to surgery. Immunohistochemistry will be performed and inflammatory invasion of the tumor will be evaluated according to Klintrup's methods (12) and the immunoscore (13). These methods are based on a scoring system defining the deepest point of invasion of inflammatory cells identified from haematoxylin and eosin slides.

Methods

Whole blood gene expression profiling:

Blood samples will be collected in PAX-gene tubes and sent for analysis at Odense University Hospital, Dept. of Clinical Genetics. Total RNA will be extracted using the Paxgene Blood RNA kit (Qiagen, Franklin Lakes, NJ, USA) and quality of RNA will be tested using Agilent 2100 Bioanalyzer (Agilent Technologies, Palo Alto, CA). The Message-AmpTM III RNA amplification kit (Ambion, Austin, TX) will be used to convert total RNA to biotin-labeled aRNA. Labeled aRNA will be hybridized to Affymetrix HGU133 Plus 2.0 chips. Data pre-processing will be done in R environment using robust multi-array average expression measure (rma) to perform background correction, normalization, and expression index calculation of all microarrays. Further high level analysis will include advanced methods for high dimensional data including supervised and unsupervised methods. Fold changes will be calculated and Significance analysis of Microarray (SAM) and t-test will be used to identify differentially expressed genes, samples and correction for multiple hypothesis testing will be performed using FDR method. Pathway analysis will be applied to identify the biological mechanisms activated by the surgical manipulation, using Gene Set Enrichment Analysis (GSEA, Broad Institute).

Assessement of inflammatory and immunological markers:

When all samples have been collected, part of the bio-banked plasma and serum will be used for measurement of concentrations of TNFα, IL-1b, IL-2, IL-6, IL-10, VEGF, TGFβ and HLA-G by ELISAs on a BEP2000 ELISA instrument (Siemens Healthcare, Erlangen, Germany) at Roskilde Hospitals, Dept.of Clinical Biochemistry, where they have a lot of experience with these measures.

Analysis of lekocyte subpopulations:

Multi-color immunophenotyping of leukocyte sub-populations will be performed within 1-2 hours after blood samples have been drawn. Analysis will be done by the use of BD FACS Canto II instruments (BD Biosciences, New Jersey, USA). This instrument analyzes eight colors/markers per tube. By the use of specific marker panels CD3+CD4+, CD3+CD8+, FoxP3+ / CD4+CD25+CD127 /dim regulatory T cells, CD4+HLA-G+ regulatory T cells, myeloid-derived suppressor cells and NK subsets will be identified. Results will be analyzed according to inflammatory and immunological up or down regulation in the period from the day before surgery and up to 10 days after.

Immunohistochemical analysis of tumor specimens:

Immunohistochemistry will be performed when all samples have been collected. Depths of invasion and number of cells expressing CD4, CD8, CD45RO and GZMB will be analyzed. The analysis will be performed according to the Klintrup's methods, which is a scoring method ranging from 0-3. A score of 0 indicates no increase in the inflammatory cells at the deepest point of the tumors invasive margin; 1 indicates a mild and patchy increase; 2 indicates a prominent inflammatory reaction, and 3 denotes a florid cup-like inflammatory infiltrate at the invasive edge with frequent destruction of cancer cell islands. These scores are then classified as low (0 and 1) and high (2 and 3) grade.

NK cells After isolation af cryopreservation of PBMC's, the functional activity of NK cells is determined in vitro by exposing them to chromium labeled NK sensitive target cells. NK cell activity is quantified in this assay by the measurement of chromium released from NK cell lysed targets.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 to 75 years of age
2. Patients diagnosed with colon cancer (UICC stadium II-III) and scheduled for laparoscopic hemicolectomy.
3. ASA class I-III (Classification of the American Society of Anesthesiology)
4. Signed informed consent

Exclusion Criteria:

1. Known immune-defects
2. Withdrawal of informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients undergoing elective, laparoscopic hemicholectomy for Colon cancer UICC stadium II-III.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Oxidative and immunological gene-expression before and after laparoscopic surgery for colon cancer using whole blood gene expression profiling from blood samples | 1 year
  The most significantly differentially expressed probe sets will be chosen for further analysis. Examples of exact genes will be genes encoding for TNFα, IL-1b, IL-2, IL-6, IL-10, VEGF, TGFβ and HLA-G. Within oxidative and antioxidative genes, special emphasis will be taken in FoxO3, TP53 and ATM.

SECONDARY OUTCOMES:
Specific immune modulating proteins in blood before and after laparoscopic surgery for colon cancer, using flow cytometry and NK-cell isolation from blood samples | 1 year
  TNFα, IL-1b, IL-2, IL-6, IL-10, VEGF, TGFβ and HLA-G, the functional activity of NK-cells, and the fractions and absolute numbers of specific sub-populations of CD3+CD4+, CD3+CD8+, FoxP3+ / CD4+CD25+CD127 /dim regulatory T cells, CD4+HLA-G+ regulatory T cells, myeloid-derived suppressor cells and NK subsets will be identified before and after surgery.
Assessement of inflammatory tumor invasion using immunohistochemestry on tumor tissue samples | 1 year
  Tumor samples will be analyzed for level of invasion of immunological cells through immunohistrochemistry and definition of the deepest point of invasion of immunological cells according to the Klinstrups methods. The results will be correlated to the results from gene expression profiling and analysis of inflammatory and immune modulating proteins determined before surgery.

IPD SHARING:
Plan to Share IPD: No